CLINICAL TRIAL: NCT05916079
Title: Breastfeeding Failure: Influence of Smartphone Use and Distraction Factors
Acronym: BRIEFCALL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2023_843_0061
Record Dates: First submitted 2023-06-13; First posted 2023-06-23 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Breastfeeding; Smartphone
Keywords: Breastfeeding; smartphone; screen; distraction; developmental care
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- breastfeeding success (Yes): Mothers are to be contacted at 1 month to assess the main outcome: breastfeeding status (Yes vs No) classified as breastfeeding success (Yes) or breastfeeding failure (No).
- breastfeeding failure (No): Mothers are to be contacted at 1 month to assess the main outcome: breastfeeding status (Yes vs No) classified as breastfeeding success (Yes) or breastfeeding failure (No).

SUMMARY:
The benefits of breastfeeding no longer need to be proven. Many studies have shown its positives effects on both infants and mothers. Exclusive breastfeeding is thus recommended within the first six months of life.

Excessive screen use has been shown to be harmful in many aspects of daily life. The impact upon the relation between mother and newborn infant is poorly studied.

The study aims to evaluate the impact of the use of smartphones on the success and duration of breastfeeding.

ELIGIBILITY:
Inclusion Criteria:

* breastfeeding mothers of Newborn breastfed infant born in the maternity ward of the Amiens-Picardie University Hospital

Exclusion Criteria:

* Mother refusing to participate in the study; hospitalization during the neonatal period

Min Age: 18 Months | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — breastfeeding mothers of Newborn infant
Study Population: breastfeeding mothers of Newborn breastfed infant born in the maternity ward of the Amiens-Picardie University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Variation of Breastfeeding status in both groups | at 2 months
  At 2 months after birth, mothers will be contacted to record their breastfeeding status.
Variation of Breastfeeding status in both groups | at 3 months
  At 3 months after birth, mothers will be contacted to record their breastfeeding status.
Variation of Breastfeeding status in both groups | at 4 months
  At 4 months after birth, mothers will be contacted to record their breastfeeding status.
Variation of Breastfeeding status in both groups | at 6 months
  At 6 months after birth, mothers will be contacted to record their breastfeeding status.

CONTACTS AND LOCATIONS:
Locations (1):
- Amiens University Hospital, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No